CLINICAL TRIAL: NCT03659292
Title: Effects of Epidural Block on the Prognosis in Patients With Pancreatic Cancer Undergoing Distal Pancreatectomy----A Multi-center Randomized Controlled Trial
Brief Title: Effects of Epidural Block on the Prognosis in Patients With Pancreatic Cancer Undergoing Distal Pancreatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Changhong Miao, Director of Anesthesiology Department of Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FDUSCCA-2
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Cancer of Pancreas
Keywords: Epidural block; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Anesthesia, Epidural; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEA+PCEA (Experimental): General anesthesia combined with epidural anesthesia will be performed during surgery and patient-controlled epidural analgesia (PCEA) will be provided after surgery.
  Interventions: Other: GEA; Other: PCEA
- GA+PCIA (Other): General anesthesia will be performed during surgery and patient-controlled intravenous analgesia (PCIA) will be provided after surgery.
  Interventions: Other: GA; Other: PCIA

INTERVENTIONS:
Other: GEA — Thoracic epidural catheterization will be performed and epidural anesthesia will be maintained with 0.25% ropivacaine during surgery. General anesthesia will be maintained with inhalation (sevoflurane) and muscle relaxants will be administered when considered necessary.
  Other Names: General anesthesia combined with epidural anesthesia
  Arms: GEA+PCEA
Other: PCEA — Patient-controlled epidural analgesia (0.15% ropivacaine and 0.5ug/ml sufentanil infusion) will be provided after surgery.
  Other Names: Patient-controlled epidural analgesia
  Arms: GEA+PCEA
Other: GA — General anesthesia will be maintained with inhalation (sevoflurane) and sufentanil infusion, and muscle relaxants will be administered when considered necessary.
  Other Names: General anesthesia
  Arms: GA+PCIA
Other: PCIA — Patient-controlled intravenous analgesia (1ug/ml sufentanil) will be provided after surgery.
  Other Names: Patient-controlled intravenous analgesia
  Arms: GA+PCIA

SUMMARY:
The purpose of this randomized controlled clinical trial is to investigate the effects of epidural block on overall survival，disease-free survival and recovery in patients with pancreatic cancer undergoing distal pancreatectomy. This study will also evaluate the effects of this technique on neuroendocrine, stress and inflammatory response in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective distal pancreatectomy for pancreatic cancer .
2. ASA statusⅠ-Ⅲ.
3. 18 years to 80 years （adults）.
4. Able to understand, communicate and sign an informed consent form.

Exclusion Criteria:

1. Laparoscopic surgery.
2. Preoperative chemotherapy or radiotherapy.
3. Pregnancy.
4. Allergic to any drugs used during the study.
5. Long-term receiving β-blockers.
6. Complicated with chronic inflammatory diseases, autoimmune diseases, or long-term receiving glucocorticoids or other immunosuppressants before surgery.
7. Abnormal coagulation functions (platelet count prior to surgery <100000/ μL , APTT value is more than the normal value, INR > 1.3 or clopidogrel that cannot be discontinued 7 days prior to surgery).
8. Complicated with severe heart disease (NYHA classification >3), severe renal insufficiency (serum creatinine >1.8mg/dL or receiving renal replacement therapy), severe hepatic disease (Child-Pugh classification=C), diabetes (fasting blood glucose not in the range of 3.9-13.8 mmol/L ), or acute infectious diseases (WBC>10000/μL) before surgery.
9. BMI > 35.
10. All contraindications to epidural block.
11. Chronic opiate medication/drug abuse.
12. Complicated with severe mental illness, cognitive disorder or unable to collaborate during the study.
13. Refuse to sign an informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | During 2 years after surgery
  Defined and calculated as the time from the date of surgery to death related to all reasons

SECONDARY OUTCOMES:
Disease-free survival (DFS ) | During 2 years after surgery
  Defined and calculated as the time from the date of surgery to the first time of pancreatic cancer recurrence or metastasis or cancer-related death
Postoperative pain score and side effects of patient-controlled analgesia | During the first 48 hours after surgery
  Assessed with visual analogue score ( 0 is no pain and 10 is the most severe pain)
Incidence of delirium | During the first 1 week after surgery
  Assessed for delirium using the 3D-CAM instrument
Incidence of persistent post-surgical pain (PPSP) after surgery | During 2 years after surgery
  Assessed with visual analogue score ( 0 is no pain and 10 is the most severe pain)
Length of stay in hospital after surgery | During the first 30 days after surgery
Return of bowel function | During the first 30 days after surgery
  Measured by the time of first flatus
Removal of Perianastomotic drains | During the first 30 days after surgery
Removal of Urinary drainage | During the first 30 days after surgery
Removal of nasogastric tube | During the first 30 days after surgery
Blood level of neuroendocrine, stress and inflammatory response | During surgery and the first 24 hours after surgery
  Changes of blood epinephrine, norepinephrine, cortisol, VEGF, interleukin-6 (IL-6)、interleukin-8 (IL-8), peripheral blood NLR ( neutrophil-lymphocyte ratio)
Blood CA19-9 、CA125、CEA、CA72-4、CA242、AFP、CA15-3、CA50 levels | During 2 years after surgery
Blood levels of ropivacaine and sufentanil | During surgery and the first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Changhong Miao, Principal Investigator — Fudan University; Qianjin Liu, Study Director — Washington University School of Medicine
Locations (3):
- China (3):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Fudan University Huashan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No